CLINICAL TRIAL: NCT07371507
Title: Effect of a Health Education Program on Teachers' Antibiotic Use Practices and Resistance Prevention: A Randomized Controlled Trial Among High School Teachers in Koya District, Iraq
Brief Title: Effect of a Health Education Program on Teachers' Antibiotic Use Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Choman Abdulqahar Khudhur, Assistant Lecturer / Researcher, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HMU-AR-TEACHERS-RCT-2026; HMU-CON-ETH-249-2024 (Other: College of Nursing, Hawler Medical University, Erbil, Iraq)
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Antibiotic Resistance Prevention
Keywords: Antibiotic Resistance; Health Education; Teachers; Antibiotic Use Practices; Randomized Controlled Trial; School-Based Intervention; Behavioral Intervention
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: Eligible teachers were individually randomized in a 1:1 ratio to either an intervention group receiving a structured health education program or a control group receiving no intervention during the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this arm received a structured health education program focused on appropriate antibiotic use, completion of prescribed treatment courses, avoidance of self-medication, and prevention of bacterial antibiotic resistance.
  Interventions: Other: Behavioral
- Control Group (No Intervention): Participants in this arm did not receive the health education intervention during the study period and continued their usual practices without additional educational input.

INTERVENTIONS:
Other: Behavioral — A structured health education program delivered to high school teachers, focusing on appropriate antibiotic use, risks of antibiotic misuse, completion of prescribed treatment courses, avoidance of self-medication, and prevention of bacterial antibiotic resistance. The program was delivered through interactive educational sessions supported by informational materials.
  Other Name: Health Education Program on Antibiotic Use and Resistance
  Other Names: Health Education Program on Antibiotic Use and Resistance
  Arms: Intervention Group

SUMMARY:
Antibiotic resistance is a growing public health problem caused in part by inappropriate use of antibiotics. Teachers play an important role in shaping health knowledge and behaviors within schools and communities. This study evaluates the effect of a structured health education program on teachers' antibiotic use practices among high school teachers in the Koya District, Erbil City, Iraq.

In this randomized controlled trial, eligible teachers were assigned to either an intervention group that received a targeted health education program on appropriate antibiotic use and resistance prevention, or a control group that did not receive the program during the study period. Teachers' antibiotic use practices were assessed before and after the intervention using a structured questionnaire.

The goal of this study is to determine whether a health education program can improve responsible antibiotic use practices and reduce behaviors that contribute to antibiotic resistance. The findings may help inform future school-based health education strategies aimed at preventing antibiotic resistance at the community level.

DETAILED DESCRIPTION:
Bacterial antibiotic resistance represents a major global health challenge driven largely by inappropriate antibiotic use, including self-medication, incomplete treatment courses, and misuse for non-bacterial illnesses. Educational interventions targeting key community members have been recognized as an effective strategy for promoting responsible antibiotic use. Teachers, as trusted role models, have the potential to influence health behaviors among students, families, and the broader community.

This study was designed as a pragmatic, individually randomized controlled trial to evaluate the effect of a health education program on teachers' antibiotic use practices among high school teachers in the Koya District, Erbil City, Iraq. Ten high schools were selected using a convenience sampling approach to ensure geographic representation across the district. Eligible teachers who consented to participate were randomly assigned in a 1:1 ratio to either an intervention group or a control group using a lottery-based randomization method.

The intervention consisted of a structured health education program focusing on appropriate antibiotic use, completion of prescribed treatment courses, avoidance of self-medication, and prevention of antibiotic resistance. The control group did not receive the educational program during the study period. Teachers' practices related to antibiotic use were assessed at baseline and after completion of the intervention using a validated questionnaire.

The primary outcome of the study was the change in antibiotic use practice scores from pre-intervention to post-intervention. Secondary outcomes included changes in knowledge and attitudes related to antibiotic use and resistance. Statistical analyses were conducted to compare outcomes between the intervention and control groups and to identify predictors of appropriate antibiotic use practices.

This trial was registered retrospectively due to delayed awareness of trial registration requirements. Participant recruitment, intervention delivery, and data collection were completed prior to registration. The authors confirm that the study protocol, outcome measures, and statistical analysis plan were not modified after data collection or analysis.

ELIGIBILITY:
Inclusion Criteria:

* High school teachers currently employed in Koya District, Erbil City, Iraq.
* Available during the study period.
* Willing to participate in the health education program and complete the study questionnaires.
* Provided written informed consent.

Exclusion Criteria:

* Teachers who previously participated in similar training programs related to antibiotic use or resistance.
* Teachers involved in the pilot study.
* Teachers who were absent during data collection periods.
* Teachers who declined participation or did not complete the pre- or post-intervention assessments.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Antibiotic Use Practice Score | From baseline (pre-intervention) to post-intervention (approximately 8 weeks)
  Change in teachers' antibiotic use practice score measured using the Antibiotic Use Practice Questionnaire, a validated 16-item self-reported scale assessing appropriate antibiotic use, completion of prescribed treatment courses, avoidance of self-medication, and behaviors related to antibiotic resistance prevention. Each item is scored on a 5-point Likert scale (1 = never to 5 = always), resulting in a total score range of 16 to 80, with higher scores indicating better and more appropriate antibiotic use practices.

CONTACTS AND LOCATIONS:
Locations (1):
- High Schools in Koya District, Erbil City, Erbil, Erbil Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. Antimicrobial resistance. Geneva: World Health Organization; 2023. Available from: https://www.who.int/news-room/fact-sheets/detail/antimicrobial-resistance